CLINICAL TRIAL: NCT03866291
Title: ESBL-producing Enterobacteriaceae in Patients With Traveller's Diarrhoea- a Prospective Cohort Study.
Brief Title: ESBL in Patients Returning to Sweden With Traveller's Diarrhoea
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0123
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Antibiotic Resistant Infection; Antibiotic Resistant Strain; Traveler's Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectal cultures and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESBL carrier: This cohort is followed for a year with additional selective ESBL cultures after 1, 3, 6 and 12 months. In the end of the year a questionnaire is handed in to the study group.
  Sera is donated after 4-6 weeks and in year.
  Interventions: Other: No intervention, observational
- Non ESBL-carrier: No further rectal cultures. In the end of the year a questionnaire is handed in to the study group. Sera is donated after 4-6 weeks and in year.
  Interventions: Other: No intervention, observational

INTERVENTIONS:
Other: No intervention, observational — See above

SUMMARY:
Patients with traveller's diarrhoea frequently harbour Extended Spectrum Betalactamase (ESBL)-producing Enterobacteriaceae (EPE) returning from EPE-endemic areas.

This study investigates to what extent travellers returning to Sweden with traveller's diarrhoea carry ESBL in their stool. The isolates are examined further according to species, phenotype, antibiogram and whole genome sequencing.

DETAILED DESCRIPTION:
Samples sent to the department of clinical microbiology in Lund, Sweden for culture of salmonella, shigella, yersinia or campylobacter are also cultured selectively for ESBL.

All patients are contacted by mail with the results. ESBL-positive patients are invited to submit further faecal cultures and blood samples during one year follow up time, to investigate how long the patient is colonized with ESBL.

ELIGIBILITY:
Inclusion Criteria:

* Travellers diarrhoea
* foreign traveller

Exclusion Criteria:

* foreign traveller but no symptoms

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Travellers of all ages
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion ESBL-colonized after one year. | 1 year
  Defined as a Positive ESBL-culture obtained 12 months after travel

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ljungquist, Principal Investigator — Lunds Universitet
Locations (1):
- Oskar Ljungquist, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ljungquist O, Camporeale A, Nematzadeh S, Giske CG, Resman F, Riesbeck K, Tham J. A Cross-Sectional Cohort Study of Extended-Spectrum-Beta-Lactamase-Producing Enterobacterales in Patients with Traveler's Diarrhea. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01585-20. doi: 10.1128/AAC.01585-20. Print 2020 Nov 17. PMID 32988817